CLINICAL TRIAL: NCT00999284
Title: Ophthalmologic Examinations After 4-hour Infusion of ZK200775 in Healthy Elder Male Volunteers
Brief Title: Ophthalmologic Examinations After Infusion of ZK200775
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Bayer (Industry)
Responsible Party: Dr. Thomas Staks, Bayer Schering Pharma AG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 96048
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2009-10-21 (Estimated); Status verified 2009-10

CONDITIONS: Visual Acuity
Keywords: ZK200775 is tested for its effects on vision on healthy probands.
MeSH Terms: interventions — ZK 200775; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Sham infusion of sodium chloride 0.9%
  Interventions: Drug: Sodium Chloride
- Low dose arm (Active Comparator): Infusion of 0.3 mg/kg/h ZK200775 over 4 hours
  Interventions: Drug: ZK200775
- High dose arm (Active Comparator): Infusion of 0.75 mg/kg/h ZK200775 over 4 hours
  Interventions: Drug: ZK200775

INTERVENTIONS:
Drug: ZK200775 — Intravenous infusion of 0.3 mg/kg/h of ZK200775 over a period of 4 hours.
  Arms: Low dose arm
Drug: ZK200775 — Intravenous infusion of 0.75 mg/kg/h of ZK200775 over a period of 4 hours.
  Arms: High dose arm
Drug: Sodium Chloride — Intravenous infusion of sodium chloride over a period of 4 hours.
  Arms: Placebo

SUMMARY:
ZK 200775 is an antagonist at the α-Amino-3-hydroxy-5-methyl-4-isoxazolepropionate (AMPA) receptor and had earned attention a possible neuroprotective agent in cerebral ischemia. Probands receiving the agent within a stroke therapy related Phase I trial reported on an alteration of visual perception. In this trial, the effects of ZK 200775 on the visual system will be analyzed in detail.

In a randomised, placebo-controlled, double-blind study eyes and vision will be examined before and after the intravenous administration of ZK 200775. The following methods will be applied: clinical examination, visual acuity, ophthalmoscopy, colour vision, rod absolute threshold, central visual field, pattern-reversal visual evoked potentials (pVEP), ON-OFF and full-field electroretinogram (ERG).

ELIGIBILITY:
Inclusion Criteria:

* The participant must be a voluntary proband
* Age between 55 and 65 years
* Body weight must not exceed the following value: Body height in cm minus 100 = body weight [kg] +/- 20%
* Male sex
* Written informed consent
* Physical examination: Probands must show normal findings without clinical relevance, mental and physical health is required;

Exclusion Criteria:

* Clinical history:

  * Substantial pre-existing medical condition
  * Known allergy to the employed effective components or galenic components
* Medicaments and drugs

  * Intake of systemically or locally acting drugs which conflict with the aim of the trial or that can influence the results (antipsychotic drugs, antidepressants, barbiturates and benzodiazepines)
  * A clinical history that hints to substance or alcohol abuse
  * Nicotine abuse of more than 10 cigarettes a day
  * Consumption of alcoholic beverages on the day prior to the examinations
  * Extreme physical stress (sports or work) within 8 days prior to the examinations
  * Blood donation within 2 months prior to the examinations
  * Relevant vaccination or stay abroad
  * Special or onesided alimentation (strict vegetarianism, low-caloric diet)
  * Simultaneous participation in another clinical trial
* Vital signs (after 3 minutes of rest)

  * Blood pressure with systolic values > 160 mmHg and / or diastolic values > 95 mmHg
  * Heart frequency: Values beyond 50-100 beats per minute
* Electrocardiogram

  * abnormal 12-channel ECG
* Laboratory findings

  * Hepatitis antigen (HBsAG), hepatitis C-antibodies or positive HIV-test
* Clinical pharmacology

  * positive drug test
  * clinically relevant abnormalities of the examined parameters
* Opinion of the investigator: when due to scientific or personal reasons or matters of compliance or safety a patient should not take part in the trial
* Opacification of optic media, retinal disease, optic nerve disease, amblyopia or color vision defects
* Status post intraocular surgery (exception: cataract surgery with implantation of a posterior chamber lens), laser coagulation
* Myopia > -5 diopters, hyperopia > +5 diopters
* Narrow angle glaucoma

Ages: 55 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 1996-12; Primary Completion 1998-04 (Actual); Study Completion 1998-04 (Actual)

PRIMARY OUTCOMES:
Visual acuity

SECONDARY OUTCOMES:
Color vision (Panel D-15 test), dark vision (adaptometer), full-field electroretinogram

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Staks, Dr., Study Director — Bayer
Locations (1):
- Charité Unviversitätsmedizin Berlin, Augenklinik Campus Virchow-Klinikum, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Bergholz R, Staks T, Ruther K. Effects of the AMPA antagonist ZK 200775 on visual function: a randomized controlled trial. PLoS One. 2010 Aug 12;5(8):e12111. doi: 10.1371/journal.pone.0012111. PMID 20711429